CLINICAL TRIAL: NCT00408824
Title: Assessment of Genetic Risk of Metabolic Syndrome in Company Employee and Making New Health Guidance Program (NGK Study)
Brief Title: Investigation of Genetic Risk of Metabolic Syndrome in Company Employee (NGK Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Other Study IDs: RIEM-G-3
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Healthy; Metabolic Syndrome X; Hyperlipidemia; Hypertension; Diabetes Mellitus
Keywords: insulin resistance; adipocytokine; Metabolic syndrome; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias; Hypertension; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The metabolic syndrome is a highly prevalent disorder, which causes atherosclerotic cardiovascular disease and is closely associated with insulin resistance. The alteration of the secretion of adipocytokines from accumulated visceral adipose tissue in the obese induces insulin resistance. The purpose of this study is to identify gene polymorphisms that confer susceptibility to the metabolic syndrome and to make up a new health guidance program based on genetic risk assessment. About 25% of male employees over 45 years old in a certain company are diagnosed with the metabolic syndrome in medical examination. We, the researchers at Nagoya University, will analyze gene polymorphism and various biomarkers of over 3500 company employees.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who work for a certain company

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Yasui, MD, PhD, Study Chair — Department of Bio-information Analysis, Research Institute of Environmental Medicine, Nagoya University
Locations (1):
- Department of Bio-information Analysis, Research Institute of Environmental Medicine, Nagoya University, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Tanimura D, Shibata R, Izawa H, Hirashiki A, Asano H, Murase Y, Miyata S, Nakatochi M, Ouchi N, Ichihara S, Yasui K, Yoshida T, Naruse K, Matsubara T, Yokota M. Relation of a common variant of the adiponectin gene to serum adiponectin concentration and metabolic traits in an aged Japanese population. Eur J Hum Genet. 2011 Mar;19(3):262-9. doi: 10.1038/ejhg.2010.201. Epub 2010 Dec 8. PMID 21150884